CLINICAL TRIAL: NCT03026413
Title: The Comparison Between the Pulmonary Vein Antrum Modification by SmartTouch Ablation Catheter With Contact Force Monitoring and Circumferential Pulmonary Vein Isolation by That Without Contact Force Monitoring Plus Lasso Catheter for the Patients of Paroxysmal Atrial Fibrillation: a Randomized Controlled Trial
Brief Title: The Comparison Between the PVAM and CPVI for the Patients of PAF
Acronym: FORCE-PVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Minglong Chen, Professor and Director of Cardiac EP Vice Director of Dept. of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NJ01
Record Dates: First submitted 2016-12-27; First posted 2017-01-20 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Atrial Fibrillation; Pulmonary Vein Isolation
Keywords: atrial fibrillation; pulmonary vein isolation; Contact Force; antrum
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PVAM (Experimental): pulomonary vein antrum modification with contact force monitoring for AF
  Interventions: Procedure: pulmonary vein antrum modification
- Control arm (Active Comparator): pulmonary vein isolation without contact force
  Interventions: Procedure: pulmonary vein antrum modification

INTERVENTIONS:
Procedure: pulmonary vein antrum modification

SUMMARY:
To compare the efficacy and safety of circumferential pulmonary vein isolation without contact force with the pulmonary vein antrum modification for patients of paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
This is a single centre, prospective control study. The study will enroll 180 patients with 2:1 grouped.

ELIGIBILITY:
Inclusion Criteria:

* patients with paroxysmal atrial fibrillation refractory to drugs
* with consent

Exclusion Criteria:

* LVEF<50%
* history of cardiac surgery
* valvular heart disease
* abnormal thyroid function
* left atrial thrombus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
any recorded atrial arrhythmias proved by 7-day holter | at least 18 months follow up
  sustained at least 30s

SECONDARY OUTCOMES:
procedure time | time during patient enrollment
  time that the patient spend in the procedure room
x ray time | time during patient enrollment
  x ray spent during the procedure
adverse event | at least 18 months follow up

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neuzil P, Reddy VY, Kautzner J, Petru J, Wichterle D, Shah D, Lambert H, Yulzari A, Wissner E, Kuck KH. Electrical reconnection after pulmonary vein isolation is contingent on contact force during initial treatment: results from the EFFICAS I study. Circ Arrhythm Electrophysiol. 2013 Apr;6(2):327-33. doi: 10.1161/CIRCEP.113.000374. Epub 2013 Mar 20. PMID 23515263
- [Result] Reddy VY, Shah D, Kautzner J, Schmidt B, Saoudi N, Herrera C, Jais P, Hindricks G, Peichl P, Yulzari A, Lambert H, Neuzil P, Natale A, Kuck KH. The relationship between contact force and clinical outcome during radiofrequency catheter ablation of atrial fibrillation in the TOCCATA study. Heart Rhythm. 2012 Nov;9(11):1789-95. doi: 10.1016/j.hrthm.2012.07.016. Epub 2012 Jul 20. PMID 22820056
- See also: an article about the contact force role in ablation for AF — https://www.ncbi.nlm.nih.gov/pubmed/22820056